CLINICAL TRIAL: NCT05994846
Title: The Reynolds Innovative Spinal Electrical Stimulation Program: Transcutaneous Stimulation (RISES-T 2.0)
Brief Title: Non-Invasive Electrical and Magnetic Neuromodulation in Persons With Chronic Spinal
Acronym: RISES-T2
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding.
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Mijail Demian Serruya, Associate Professor, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Rises-T 2.0 iRISID-2023-2024
Record Dates: First submitted 2023-07-28; First posted 2023-08-16 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: Spinal Cord Injuries; Spinal Electrical Stimulation; Transcutaneous Spinal Stimulation; Transcutaneous Magnetic Simulation; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, unblinded, feasibility study where participants will serve as their own controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Experimental Treatment Arm (Experimental): Participants will receive closed-loop transcutaneous spinal cord stimulation via the RISES-T System while completing repetitive task practice
  Interventions: Device: RISES-T System

INTERVENTIONS:
Device: RISES-T System — The RISES-T system is a hardware and software platform that has been designed and developed to help people living with movement impairment due to Spinal Cord Injury (SCI) to improve and/or restore mobility. The hardware consists of a functional electrical stimulation device that delivers stimulation to the skin through surface electrodes; a series of wearable sensors that collect kinematic (IMU) data and muscle activity (EMG) data, and RISES Software, which incorporates algorithms that utilizes the streaming IMU and EMG sensor data to inform the electrical stimulation parameters and enables real-time visualization of the sensor data and stimulation parameters via Graphical User Interface (GUI).
  Other Names: Trancutaneous spinal stimulation

SUMMARY:
The objectives of this study are to (1) determine the effects of neuromodulation techniques on mobility in persons with chronic SCI, as measured by subjective and objective measures, and (2) to determine the optimal combination of techniques that modify mobility and movement in an individual. The neuromodulation techniques explored will be methods of electromagnetic stimulation - that is, electrical stimulation and magnetic stimulation.

DETAILED DESCRIPTION:
The study is designed in two Parts. Part 1 of the study will collect information about the participant's baseline mobility and muscular activation potential. The information collected in these sessions will, in effect, assess the participant's eligibility to continue in the study and move onto Part 2.

Part 1- Assessment Sessions This part of the study designed to determine (1) which, if any, of the participant's muscles respond to stimulation and, if there are responses observed, (2) what stimulation parameters and modalities would be best suited for the participant during Part 2 of the trial. The team will create a participant-specific menu of modalities and pre-defined parameters for electromagnetic stimulation (e.g., amplitude, channels, frequencies, electrode placement, etc.) from which they will select for participant visits in Part 2 of the study. They will also capture the participant's Movement Signature (the pattern of movement as measured by accelerometers and surface EMG that a person exhibits while sitting/standing at rest and/or doing specific tasks to inform Part 2 of the study. Finally, the participants will complete a Baseline Clinical Outcome Measures validated for SCI to provide baseline data prior to the neuromodulation intervention.

Part 2 - The Experimental Cycles This part of the study will consist of Intervention Sessions, in which the team will apply transcutaneous stimulation to the participant's target muscles identified in Part 1, using the parameters and modalities deemed best suited for the participant. during tasks and activities deemed most appropriate for the targeted muscles. The team will measure the effects of electromagnetic stimulation on the participant's muscle activity and movement.

The Cycle will also include Biometric sessions, where the participant will engage in a series of upper extremity, trunk and/or lower extremity repetitive tasks from their prescribed "activity library" that was created for them during Part 1 of the study and the team will measure changes in muscle tone, strength, and movement before and after stimulation. In other sessions, the participant will undergo a series of more targeted tasks with and without electromagnetic stimulation applied, to measure changes in the participant's neurophysiology, kinetics, and kinematics due to electromagnetic stimulation.

After a series of Intervention and Biometrics Sessions, if there are no changes observed in the participant's kinematics or EMG signals in the and/or in select outcome measures, the participant will enter a Parameter Optimization Session. During this session, the study team will revisit the library of stimulation parameters that were defined for the participant during Part 1 of the study and refine the parameters for use in the next Experimental Cycle. The manipulation and refinement of these parameters will be done with the aim of achieving changes in the subsequent Experimental Cycle.

The participant will continue in the study until the time that there is no observed effect of stimulation for three (3) consecutive Experimental Cycles, or may continue for a maximum of six (6) Experimental Cycles. At the end of the study, the participant will repeat the series of Clinical Outcome Measures that were completed at Baseline.

ELIGIBILITY:
Inclusion Criteria:

Has a non-progressive or central cord spinal cord injury

American Spinal Injury Association (ASIA) Impairment Scale (AIS) classification A, B, C, or D

Can participate in physical and occupational therapy rehabilitation programs

Is at minimum 12 months post-injury

Can provide informed consent

Has adequate caregiver support to facilitate participation in study

Is willing to undergo audio-visual recording sessions

-

Exclusion Criteria:

Has uncontrolled cardiopulmonary disease or cardiac symptoms (as determined by investigators)

Has any unstable or significant medical condition that is likely to interfere with study procedures or likely to confound study endpoint evaluations like severe neuropathic pain, depression, mood disorders or other cognitive disorders

Has autonomic dysreflexia that is severe, unstable, and uncontrolled or uncontrolled orthostatic hypotension that may interfere with rehabilitation.

Requires ventilator support Has an autoimmune etiology of spinal cord dysfunction/injury

Has spasms that limit the ability to participate in the study training (as determined by the Investigator)

Has skin breakdown in area(s) that will come into contact with electrodes

Has any active implanted medical device (e.g., cochlear implant, pacemaker, neurostimulator or medication infusion device) Is pregnant, planning to become pregnant or currently breastfeeding

Has concurrent participation in another drug or device trial that may interfere with this study

Has other traumatic injuries such as peripheral nerve injuries, severe musculoskeletal injuries (e.g., shattered pelvis, long bone fractures), that prevent evaluation of response to or participation in rehabilitation.

Is not a candidate for other reason determined by the investigators

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Spinal Cord Injury-Motor Index (SCI MovIN) | Starting 4 weeks after consent, 3 times every 2 weeks for up to 22 weeks
  evaluates movement, and recovery of neurotypical movement, within a functional context that accounts for compensations and disallows substitutions
Modified Ashworth Scale (MAS) | Starting 4 weeks after consent, 3 times every 2 weeks for up to 22 weeks
  measures spasticity in patients with lesions to the central nervous system. MAS is an assessment that is used to measure the increase in muscle tone
Manual Muscle Testing (MMT) | Starting 4 weeks after consent, 3 times every 2 weeks for up to 22 weeks
  standardized set of assessments that measure muscle strength and function

SECONDARY OUTCOMES:
Capabilities of Upper Extremity Test (CUE-T) | Once at 2 weeks after consent, and once within 9-24 weeks after consent
  A performance measure intended to assess upper extremity function following spinal cord injury (SCI)
PROMIS Pain Interference- Adult Short Form 8a (PROMIS-PI) | Once at 2 weeks after consent, and once within 9-24 weeks after consent
  A patient self-reported measure of consequences of pain on aspects of their life
Walking Index for SCI (WISCI-II) | Once at 2 weeks after consent, and once within 9-24 weeks after consent
  A measure of physical assistance needed, as well as devices required, for walking following paralysis that results from SCI
Numeric Pain Rating Scale (NPRS) | Once at 2 weeks after consent, and once within 9-24 weeks after consent
  The patient reported outcome measure the subjective intensity of pain
Patient Global Impression of Change (PGIC) Questionnaires (bowel program, bladder function, dysreflexia, pain, sensation) | Once at 2 weeks after consent, and once within 9-24 weeks after consent
  Questionnaires to assess the status of or changes in bladder function, bowel regimen, dysreflexia, pain and sensation.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerasimenko Y, Gorodnichev R, Moshonkina T, Sayenko D, Gad P, Reggie Edgerton V. Transcutaneous electrical spinal-cord stimulation in humans. Ann Phys Rehabil Med. 2015 Sep;58(4):225-231. doi: 10.1016/j.rehab.2015.05.003. Epub 2015 Jul 20. PMID 26205686
- [Background] Manson G, Atkinson DA, Shi Z, Sheynin J, Karmonik C, Markley RL, Sayenko DG. Transcutaneous spinal stimulation alters cortical and subcortical activation patterns during mimicked-standing: A proof-of-concept fMRI study. Neuroimage Rep. 2022 Jun;2(2):100090. doi: 10.1016/j.ynirp.2022.100090. Epub 2022 Mar 8. PMID 36212800
- [Background] Kumru H, Rodriguez-Canon M, Edgerton VR, Garcia L, Flores A, Soriano I, Opisso E, Gerasimenko Y, Navarro X, Garcia-Alias G, Vidal J. Transcutaneous Electrical Neuromodulation of the Cervical Spinal Cord Depends Both on the Stimulation Intensity and the Degree of Voluntary Activity for Training. A Pilot Study. J Clin Med. 2021 Jul 25;10(15):3278. doi: 10.3390/jcm10153278. PMID 34362062
- [Background] Rejc E, Smith AC, Weber KA 2nd, Ugiliweneza B, Bert RJ, Negahdar M, Boakye M, Harkema SJ, Angeli CA. Spinal Cord Imaging Markers and Recovery of Volitional Leg Movement With Spinal Cord Epidural Stimulation in Individuals With Clinically Motor Complete Spinal Cord Injury. Front Syst Neurosci. 2020 Oct 21;14:559313. doi: 10.3389/fnsys.2020.559313. eCollection 2020. PMID 33192348
- [Background] Barss TS, Parhizi B, Porter J, Mushahwar VK. Neural Substrates of Transcutaneous Spinal Cord Stimulation: Neuromodulation across Multiple Segments of the Spinal Cord. J Clin Med. 2022 Jan 27;11(3):639. doi: 10.3390/jcm11030639. PMID 35160091
- [Background] Capogrosso M, Wagner FB, Gandar J, Moraud EM, Wenger N, Milekovic T, Shkorbatova P, Pavlova N, Musienko P, Bezard E, Bloch J, Courtine G. Configuration of electrical spinal cord stimulation through real-time processing of gait kinematics. Nat Protoc. 2018 Sep;13(9):2031-2061. doi: 10.1038/s41596-018-0030-9. PMID 30190556
- [Background] Wenger N, Moraud EM, Gandar J, Musienko P, Capogrosso M, Baud L, Le Goff CG, Barraud Q, Pavlova N, Dominici N, Minev IR, Asboth L, Hirsch A, Duis S, Kreider J, Mortera A, Haverbeck O, Kraus S, Schmitz F, DiGiovanna J, van den Brand R, Bloch J, Detemple P, Lacour SP, Bezard E, Micera S, Courtine G. Spatiotemporal neuromodulation therapies engaging muscle synergies improve motor control after spinal cord injury. Nat Med. 2016 Feb;22(2):138-45. doi: 10.1038/nm.4025. Epub 2016 Jan 18. PMID 26779815
- [Background] Najib U, Bashir S, Edwards D, Rotenberg A, Pascual-Leone A. Transcranial brain stimulation: clinical applications and future directions. Neurosurg Clin N Am. 2011 Apr;22(2):233-51, ix. doi: 10.1016/j.nec.2011.01.002. PMID 21435574
- [Background] Pascual-Leone A, Freitas C, Oberman L, Horvath JC, Halko M, Eldaief M, Bashir S, Vernet M, Shafi M, Westover B, Vahabzadeh-Hagh AM, Rotenberg A. Characterizing brain cortical plasticity and network dynamics across the age-span in health and disease with TMS-EEG and TMS-fMRI. Brain Topogr. 2011 Oct;24(3-4):302-15. doi: 10.1007/s10548-011-0196-8. Epub 2011 Aug 14. PMID 21842407
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552